CLINICAL TRIAL: NCT00348556
Title: Efficacy of Intra-renal Infusion of BNP in Enhancing Renal Function in Human CHF With Cardiorenal Syndrome: A Pilot Study
Brief Title: Use of Nesiritide (BNP) in Kidney Function in Patients With Congestive Heart Failure (CHF) and Kidney Failure
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company providing catheter bought out, funding and supplies terminated
Sponsor: Horng Chen (Other)
Collaborators: FlowMedica, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Horng Chen, MD, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-004007
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2012-10-17 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Cardiorenal Syndrome
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nesiritide (Experimental): Subjects received an intrarenal infusion of nesiritide at 0.005 microgram/kg/min for 6 hours, 0.01 microgram/kg/min for 6 hours, 0.02 microgram/kg/min for 6 hours, and 0.03 microgram/kg/min for 6 hours.
  Interventions: Drug: Nesiritide

INTERVENTIONS:
Drug: Nesiritide — Nesiritide 0.005 ug/kg/min IV for 6 hours, then to 0.01 ug/kg/min for 6 hours then to 0.02ug/kg/min for 6 hours then to 0.03 ug/kg/min for the last 6 hours.
  Other Names: Natrecor; brain natriuretic peptide (BNP)

SUMMARY:
The objective of this study is to determine the safety and effectiveness of intrarenal administration of brain natriuretic peptide (BNP) in improving renal function as measured by glomerular filtration rate (GFR) and sodium excretion in patients hospitalized with acute congestive heart failure (CHF) and deterioration of kidney function (cardiorenal syndrome).

ELIGIBILITY:
Inclusion Criteria

* Age 18 years and older
* Clinical diagnosis of class III-IV CHF requiring hospitalization
* Current acute CHF decompensation
* Systolic BP > 90 mmHg
* Stable cardiac rhythm
* Estimated creatinine clearance by the Cockcroft-Gault equation of less than or equal to 60 mL/min.
* Worsening renal function after greater than or equal to 24 hours of standard therapy as defined by a plasma creatinine concentration greater than their admission of 0.3 mg/dL and a 10% increase from hospital admission creatinine OR creatinine which remains at 0.3 mg/dL and 10% increase from baseline draw done within 4 weeks of hospitalization
* Ability to provide informed consent

Exclusion Criteria

* Patients needing emergency coronary revascularization or those who may have rapidly changing cardiac function (i.e., patients with acute myocardial infarction or shock)
* Peritoneal or hemodialysis within 90 days or anticipation that dialysis or ultrafiltration of any form will be required during the study period
* Systolic blood pressure < 90 mmHg or cardiogenic shock
* Requirement of pressors for maintenance of blood pressure
* Intra-aortic blood pump use
* History of significant uncorrected renal artery stenosis as defined by >50% stenosis
* Severe aortic or mitral stenosis or significant LV outflow tract obstruction
* Pregnant or nursing women
* Prisoners
* Contraindication to nesiritide
* Contraindication to heparin
* Cause of acute renal dysfunction can be reasonably ascribed to factors other than heart failure or its treatment
* Inability to have NSAID dose held for up to 30 hours, if being treated with these medications
* Ongoing treatment with calcineurin inhibitors (cyclosporine or tacrolimus)
* Administration of radiocontrast medium within 7 days of enrollment or anticipated use of such agents during the study (other than the minimal contrast required to place the renal infusion catheter)
* Known bleeding diathesis
* Known condition that would increase the likelihood of vascular perforation or trauma, dissection such as Marfan's syndrome, cystic medial necrosis, abdominal or thoracoabdominal aortic dissection, mycotic aneurysm, abdominal aneurysm, thoracoabdominal aneurysm, renal artery aneurysm, thoracic aneurysm involving the visceral region of the aorta, and severe calcification in the area of the renal arteries
* Solitary kidney or solitary functioning kidney
* Iodine allergy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horng H. Chen, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Mayo Clinic in Rochester, MN.
Period: Overall Study
Arm/Group | Nesiritide
Started | 4
Completed | 3
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nesiritide
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Glomerular Filtration Rate (GFR) at 24 Hours
Description: Kidney function was to be measured by GFR determined by iothalamate clearance. GFR describes the flow rate of filtered fluid through the kidney measured in milliliters per minute per 1.73 m^2 of body surface area. A lower GFR means the kidney is not filtering normally. An estimated GFR of less than 60 mg/min/1.73 m^2 of body surface area is considered to be impaired kidney function.
Time Frame: baseline, 24 hours after start of infusion
Population: The data from the 3 subjects were incomplete and could not be analyzed.
Arm/Group | Nesiritide
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Urinary Sodium Excretion at 24 Hours
Description: The fractional excretion of sodium (FENa) measures the percent of filtered sodium that is excreted in the urine. This calculation is widely used to help differentiate prerenal disease (decreased renal perfusion) from acute tubular necrosis (ATN) as the cause of acute kidney injury (AKI, formerly called acute renal failure).
Time Frame: baseline, 24 hours after start of infusion
Population: The data from the 3 subjects were incomplete and could not be analyzed.
Arm/Group | Nesiritide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All adverse events that occured between enrollment in the study and 24 hours after stopping the infusion were reported.
Arm/Group | Nesiritide
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nesiritide (N=4)
Intrarenal catheter occluded (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early because the company providing catheter was bought out, and funding and supplies were terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No